CLINICAL TRIAL: NCT01731886
Title: A Randomized Clinical Trial of Lenalidomide (CC-5013) and Dexamethasone With and Without Autologous Peripheral Blood Stem Cell Transplant in Patients With Newly Diagnosed Multiple Myeloma
Brief Title: Lenalidomide and Dexamethasone With/Without Stem Cell Transplant in Patients With Multiple Myeloma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Suzanne Lentzsch, MD, Associate Clinical Professor of Clinical Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAJ2355; NCT00777881 (obsolete NCT alias)
Record Dates: First submitted 2012-11-19; First posted 2012-11-22 (Estimated); Results first posted 2019-10-15 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Multiple Myeloma
Keywords: Stem cell transplant; plasma cell myeloma; multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; Dexamethasone; Calcium Dobesilate; Hematopoietic Stem Cell Mobilization; Melphalan; Granulocyte Colony-Stimulating Factor; Filgrastim; Cyclophosphamide; Mesna

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Active Comparator): Subjects will receive the current standard of care treatment. Lenalidomide and dexamethasone for four 28-day cycles followed by steam cell collection and autologous peripheral blood stem cell transplant. After 90 days, start the maintenance phase (lenalidomide days 1-21 every 28 days for two years or until your disease progresses).
  Interventions: Procedure: Autologous peripheral blood stem cell transplant; Drug: Lenalidomide; Drug: Dexamethasone; Procedure: Stem cell collection; Drug: Melphalan; Drug: G-CSF; Drug: Cyclophosphamide; Drug: Mesna
- Arm B (Active Comparator): Subjects will receive the new treatment that will be compared with the standard of care. Lenalidomide and dexamethasone for eight 28-day cycles. After four cycles your stem cells will be collected (stem cell collection). After an additional four cycles of lenalidomide (a total of 8 cycles), start the maintenance phase (lenalidomide days 1-21 every 28 days for two years or until your disease progresses).
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone; Procedure: Stem cell collection; Drug: Cyclophosphamide; Drug: Mesna

INTERVENTIONS:
Procedure: Autologous peripheral blood stem cell transplant — Subjects deemed suitable by the principal investigator will undergo autologous peripheral blood stem cell transplantation on day 0.
  Arms: Arm A
Drug: Lenalidomide — Administered orally at a dose 25 mg daily on days 1-21 of each 28-day cycle.
  Other Names: CC-5013; Revlimid
Drug: Dexamethasone — Administered orally at a dose of 40 mg daily on days 1, 8, 15, 22 of each cycle.
  Other Names: Decadron; Hexadrol; Dexameth; Dexone; DXM
Procedure: Stem cell collection — Peripheral stem cell collection will be performed at marrow recovery, usually when white blood cell (WBC) is >2500 x 109 cells/liter; platelet count is >20 x 103/mm3.
  Other Names: Stem Cell Mobilization
Drug: Melphalan — Subjects undergoing autologous peripheral blood stem cell transplant will receive melphalan 200 mg/m2 intravenously on days -2 and -1 or only on day -2.
  Other Names: Evomela
  Arms: Arm A
Drug: G-CSF — Subjects will receive G-CSF subcutaneously daily beginning on day 5 and until blood counts recover.
  Other Names: Granulocyte-colony stimulating factor (CSF); Filgrastim
  Arms: Arm A
Drug: Cyclophosphamide — Subjects may receive up to the maximum recommended high-dose of cyclophosphamide at 4 gm/m2 intravenously.
  Other Names: Cytophosphane
Drug: Mesna — Mesna will be provided with the cyclophosphamide.
  Other Names: Mesnex

SUMMARY:
The study is being done to compare the combination of lenalidomide and dexamethasone followed by autologous peripheral blood stem cell transplant (PBSCT) and lenalidomide and dexamethasone without PBSCT in patients with untreated multiple myeloma. This comparison will include how the subjects respond to each study treatment combination, and what side effects are caused by each combination.

DETAILED DESCRIPTION:
Multiple myeloma is a malignant plasma cell proliferative disorder responsible for 11, 000 deaths each year in the United States. Approximately one third of myeloma patients develop hypercalcemia and about two thirds present with anemia. As the second most common hematologic malignancy, myeloma remains incurable. In the last forty years, options for therapy have included melphalan-prednisone, anthracyclines, and vinca alkaloids; however, relapse with those regimens continues to be inevitable with a median survival of 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed Multiple Myeloma, Salmon-Durie Stage II or III or International Staging System II or III that has not been previously treated.
* Bone marrow plasmacytosis with > or = 10% plasma cells, or sheets of plasma cells or a biopsy-proven plasmacytoma.
* Measurable levels of monoclonal protein (M protein): 1 g/dL Immunoglobulin G (IgG) or .5 g/dL Immunoglobulin A (IgA) on serum protein electrophoresis or > 200 mg of monoclonal light chain on a 24 hour urine protein electrophoresis.
* Age > or = 18 years.
* Life expectancy of greater than 12 months.
* Eastern Cooperative Oncology Group (ECOG) performance status < or = 2 (Karnofsky > or = 60%).
* Adequate organ and marrow function as defined below:

  * Hgb > or = 9 g/dL
  * Absolute Neutrophil Count > or = 1,500/ ml
  * Platelets > or = 50,000/mm3
  * Total Bilirubin < or = 1.5 mg/dL
  * Aspartate aminotransferase (AST)(SGOT) / alanine aminotransferase (ALT)(SGPT) < or = 2.5 X upper limit of normal (ULN)
  * Creatinine < 2.0 mg/dL
  * Creatinine Clearance > or = 50 ml/min
* Registered into the mandatory Revlimid REMS® program, and be willing and able to comply with the requirements of the REMS® program.
* Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid REMS® program.
* Ability to understand and the willingness to sign a written informed consent document.
* Subjects with a history of prior malignancy are eligible provided there is no active malignancy and a low expectation of recurrence within 6 months.
* Must be willing and able to take prophylaxis with either aspirin at 81 mg/day or alternative prophylaxis with either low molecular weight heparin or warfarin as recommended.
* Eligible for transplant with an age up to and including 75 years.
* Subjects in Arm A who are refusing transplant can go onto Arm B and will be evaluated separately.
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 milli-international units per millilitre (mIU/mL) within 10 - 14 days prior to and again within 24 hours of prescribing lenalidomide and must either commit to continued abstinence or 2 acceptable methods of birth control. FCBP must also agree to ongoing pregnancy testing. Males must agree to use a latex condom.

Exclusion Criteria:

* Have had chemotherapy or radiotherapy for multiple myeloma within 4 weeks of baseline.
* Receiving any other investigational agents or therapy within 28 days of baseline.
* Brain metastases.
* Subjects who are pregnant or breast feeding.
* History of previous deep vein thrombosis or pulmonary embolism must be on anticoagulation therapy with low molecular weight heparin or warfarin at therapeutic dosages (e.g. International Normalized Ratio (INR) 2-3).
* If a subject is on full-dose anticoagulants, the following criteria should be met for enrollment:

  * Must not have active bleeding or pathological conditions that carry high risk of bleeding (e.g. tumor involving major vessels, known varices).
  * Must not have thrombocytopenia requiring transfusion.
  * Must have a platelet count > 50,000.
  * Must have stable INR between 2-3.
* Smoldering myeloma or monoclonal gammopathy of undetermined significance.
* Active, uncontrolled infection.
* Active, uncontrolled seizure disorder (seizures in the last 6 months).
* Concurrent use of other anti-cancer agents or treatments.
* Positive for HIV or infectious hepatitis, type B or C.
* Hypersensitivity to thalidomide.
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2017-04-11 (Actual); Study Completion 2017-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Lentzsch, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be coded and shared with the University of Pittsburgh at the end of the trial.
Supporting Information: Study Protocol, SAP
Time Frame: After completion of the study.
Access Criteria: All data will be coded with study identifiers.

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Low-dose Dexamethasone + Stem Cell Transplantation: Subjects will receive the current standard of care treatment. Lenalidomide and dexamethasone for four 28-day cycles followed by stem cell collection and autologous peripheral blood stem cell transplant. After 90 days, start the maintenance phase (lenalidomide days 1-21 every 28 days for two years or until your disease progresses).
  Autologous peripheral blood stem cell transplant: Subjects deemed suitable by the principal investigator will undergo autologous peripheral blood stem cell transplantation on day 0.
  Lenalidomide: Administered orally at a dose 25 mg daily on days 1-21 of each 28-day cycle.
  Dexamethasone: Administered orally at a dose of 40 mg daily on days 1, 8, 15, 22 of each cycle.
  Stem cell collection: Peripheral stem cell collection will be performed at marrow recovery, usually when white blood cell (WBC) is >2500 x 109 cells/liter; platelet count is >20 x 103/mm3.
  Melphalan: Subjects undergoing autologous peripheral blood stem cell transplant will receive
- Arm B: Low-dose Dexamethasone: Subjects will receive the new treatment that will be compared with the standard of care. Lenalidomide and dexamethasone for eight 28-day cycles. After four cycles your stem cells will be collected (stem cell collection). After an additional four cycles of lenalidomide (a total of 8 cycles), start the maintenance phase (lenalidomide days 1-21 every 28 days for two years or until your disease progresses).
  Lenalidomide: Administered orally at a dose 25 mg daily on days 1-21 of each 28-day cycle.
  Dexamethasone: Administered orally at a dose of 40 mg daily on days 1, 8, 15, 22 of each cycle.
  Stem cell collection: Peripheral stem cell collection will be performed at marrow recovery, usually when white blood cell (WBC) is >2500 x 109 cells/liter; platelet count is >20 x 103/mm3.
  Cyclophosphamide: Subjects may receive up to the maximum recommended high-dose of cyclophosphamide at 4 gm/m2 intravenously.
  Mesna: Mesna will be provided with the cyclophosphamide.
Period: Overall Study
Arm/Group | Arm A: Low-dose Dexamethasone + Stem Cell Transplantation | Arm B: Low-dose Dexamethasone
Started | 31 | 29
Completed | 29 | 28
Not Completed | 2 | 1
Not completed — Death | 1 | 0
Not completed — Never started treatment | 0 | 1
Not completed — Non-compliant | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm A: Low-dose Dexamethasone + Stem Cell Transplantation: Subjects will receive the current standard of care treatment. Lenalidomide and dexamethasone for four 28-day cycles followed by stem cell collection and autologous peripheral blood stem cell transplant. After 90 days, start the maintenance phase (lenalidomide days 1-21 every 28 days for two years or until your disease progresses).
- Arm B: Low-dose Dexamethasone: Subjects will receive the new treatment that will be compared with the standard of care. Lenalidomide and dexamethasone for eight 28-day cycles. After four cycles your stem cells will be collected (stem cell collection). After an additional four cycles of lenalidomide (a total of 8 cycles), start the maintenance phase (lenalidomide days 1-21 every 28 days for two years or until your disease progresses).
- Total: Total of all reporting groups
Arm/Group | Arm A: Low-dose Dexamethasone + Stem Cell Transplantation | Arm B: Low-dose Dexamethasone | Total
Number analyzed (Participants) | 31 | 29 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 18 | 39
  >=65 years | 10 | 11 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 12 | 27
  Male | 16 | 17 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 6 | 10
  White | 23 | 20 | 43
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 3 | 3 | 6
ISS Stage [Count of Participants; unit: Participants]
  Stage 1(B2M <3.5 mg/L and serum albumin ≥3.5 g/dL) | 11 | 11 | 22
  Stage 2(Neither stage I nor stage III) | 14 | 14 | 28
  Stage 3(B2M ≥5.5 mg/L) | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate
Description: The primary objective of this study is to determine the complete response rate of lenalidomide and low-dose dexamethasone versus that of lenalidomide and low-dose dexamethasone followed by autologous peripheral blood stem cell transplant in patients with newly diagnosed multiple myeloma (will include unconfirmed complete response (CR), CR and stringent complete response (sCR)).
Time Frame: 3 years
Population: 1 participant in Arm B never started treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Low-dose Dexamethasone + Stem Cell Transplantation | Arm B: Low-dose Dexamethasone
Number analyzed (Participants) | 31 | 28
Participants | 7 | 7

2. Secondary Outcome: Overall Survival Rate (OS)
Description: To compare overall survival in subjects receiving autologous peripheral blood stem cell transplant after undergoing induction therapy with lenalidomide and dexamethasone versus in those receiving only lenalidomide and dexamethasone, followed by lenalidomide maintenance in both arms. Only patients who achieved at least a partial response (PR) following 4 cycles of induction were included in the analysis.
Time Frame: 4 years
Population: Only patients who achieved at least a partial response (PR) following 4 cycles of induction were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Arm B: Low-dose Dexamethasone: Subjects will receive the new treatment that will be compared with the standard of care. Lenalidomide and dexamethasone for eight 28-day cycles. After four cycles your stem cells will be collected (stem cell collection). After an additional four cycles of lenalidomide (a total of 8 cycles), start the maintenance phase (lenalidomide days 1-21 every 28 days for two years or until your disease progresses).
  Only includes subjects who received drug.
Arm/Group | Arm A: Low-dose Dexamethasone + Stem Cell Transplantation | Arm B: Low-dose Dexamethasone
Number analyzed (Participants) | 25 | 19
percentage of participants | 79.8 [64.0 to 95.6] | 78.9 [60.6 to 97.3]

3. Secondary Outcome: Overall Survival Rate (OS)
Description: as for outcome 2
Time Frame: 2 years
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Low-dose Dexamethasone + Stem Cell Transplantation | Arm B: Low-dose Dexamethasone
Number analyzed (Participants) | 25 | 19
percentage of participants | 100 [95 to 100] | 94.7 [85.4 to 99.9]

4. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is the length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse.
Time Frame: 4 years
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Low-dose Dexamethasone + Stem Cell Transplantation | Arm B: Low-dose Dexamethasone
Number analyzed (Participants) | 25 | 19
percentage of participants | 36.0 [17.2 to 54.8] | 31.6 [10.7 to 52.5]

5. Secondary Outcome: Progression Free Survival (PFS)
Description: as for outcome 4
Time Frame: 2 years
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Low-dose Dexamethasone + Stem Cell Transplantation | Arm B: Low-dose Dexamethasone
Number analyzed (Participants) | 25 | 19
percentage of participants | 52.0 [32.4 to 71.6] | 47.4 [24.9 to 69.8]

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Arm A: Low-dose Dexamethasone + Stem Cell Transplantation | Arm B: Low-dose Dexamethasone
All-Cause Mortality (participants affected / at risk) | 14/31 | 11/28
Serious Adverse Events (participants affected / at risk) | 7/31 | 7/28
Other Adverse Events (participants affected / at risk) | 21/31 | 19/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Low-dose Dexamethasone + Stem Cell Transplantation (N=31) | Arm B: Low-dose Dexamethasone (N=28)
Presyncope (Cardiac disorders) | 0 (0) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (2)
Febrile Neutropenia (Infections and infestations) | 1 (2) | 0 (0)
Infection with Grade 3 or 4 Neutrophils (Infections and infestations) | 1 (1) | 1 (1) — Anal/Perianal
Infection (Infections and infestations) | 0 (0) | 1 (1)
Lung Infection (Infections and infestations) | 1 (3) | 0 (0)
Myelodysplastic Syndrome (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Neoplasms (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Pain (General disorders) | 1 (2) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Abdominal Pain (General disorders) | 0 (0) | 1 (1)
Back Pain (General disorders) | 0 (0) | 1 (1)
Skin Infection (Infections and infestations) | 1 (1) | 0 (0)
Syncope (General disorders) | 1 (1) | 0 (0)
Thromboembolic Event (Vascular disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Low-dose Dexamethasone + Stem Cell Transplantation (N=31) | Arm B: Low-dose Dexamethasone (N=28)
Anemia (Blood and lymphatic system disorders) | 2 (12) | 4 (14)
Diarrhea (Gastrointestinal disorders) | 3 (7) | 5 (11)
Decreased Neutrophil Count (Blood and lymphatic system disorders) | 8 (22) | 4 (7)
Decreased WBC Count (Blood and lymphatic system disorders) | 6 (13) | 3 (7)
Decreased Platelet Count (Blood and lymphatic system disorders) | 5 (24) | 1 (1)
Abnormal Neutrophils/Granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 5 (11) | 7 (26)
Pain in extremity (General disorders) | 2 (3) | 1 (6)
Increased Alanine Aminotransferase (Hepatobiliary disorders) | 2 (6) | 2 (3)
Cough (General disorders) | 4 (7) | 3 (3)
Insomnia (General disorders) | 3 (4) | 5 (7)
Infection (Infections and infestations) | 3 (5) | 5 (7)
Abnormal Leukocytes (Blood and lymphatic system disorders) | 2 (3) | 3 (8)
Abnormal Platelet Count (Blood and lymphatic system disorders) | 2 (3) | 4 (12)
Abnormal Hemoglobin (Blood and lymphatic system disorders) | 1 (1) | 3 (8)
Upper Respiratory Infection (Infections and infestations) | 1 (2) | 2 (3)
Urinary Tract Infection (Infections and infestations) | 2 (3) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) | 3 (5)
Paresthesia (General disorders) | 0 (0) | 3 (4)
Nausea (General disorders) | 2 (3) | 2 (4)
Hyponatremia (Metabolism and nutrition disorders) | 2 (3) | 1 (2)
Fatigue (General disorders) | 3 (4) | 3 (5)
Abdominal Pain (General disorders) | 2 (4) | 1 (1)
Fever (Infections and infestations) | 1 (2) | 2 (3)
Decreased Lymphocyte Count (Blood and lymphatic system disorders) | 0 (0) | 3 (6)
Musculoskeletal and Connective Tissue Disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-19): https://cdn.clinicaltrials.gov/large-docs/86/NCT01731886/Prot_SAP_000.pdf